CLINICAL TRIAL: NCT06420323
Title: NovoX® Cup as Primary Dressing After Breast Reduction: an Intra-individual Comparison Between Standard of Care and Oxygen-enriched Olive Oil Bra Cup
Brief Title: NovoX®Cup as Primary Dressing After Breast Reduction
Status: Recruiting | Type: Observational
Sponsor: MOSS S.p.A. (Industry)
Responsible Party: Sponsor
Other Study IDs: NOVOX CUP
Record Dates: First submitted 2024-05-14; First posted 2024-05-20 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Wound Healing Disorder; Post-Surgical Complication; Mammaplasty
Keywords: Surgical wounds; Breast surgery; Plastic surgery; Oxygen-enriched oil; Dressing; Wound healing; Scar quality; postoperative complications; Breast reduction
MeSH Terms: conditions — Surgical Wound; Postoperative Complications | interventions — Therapeutics

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Treatment with NovoX® Cup: Patient gets treated with NovoX® Cup for 2 weeks.
  Interventions: Device: Treatment with NovoX® Cup
- Treatment with Omnistrip®: Patient gets treated with Omnistrip® for 2 weeks.
  Interventions: Device: Treatment with Omnistrip®

INTERVENTIONS:
Device: Treatment with NovoX® Cup — NovoX® Cup treatment
  Groups: Treatment with NovoX® Cup
Device: Treatment with Omnistrip® — Omnistrip® treatment
  Groups: Treatment with Omnistrip®

SUMMARY:
Breast reduction is one of the most frequently performed plastic surgeries. Studies have shown that breast reduction surgery significantly improves the patients' suffering and leads to a better health-related quality of life.However, as in every surgery, there can be complications. Wound disorders, such as open wounds and skin loss account for the most commonly encountered postoperative complications. NovoX® Cup is a new single-use wound dressing that is shaped cupular in order to tightly adapt to the breast anatomy. It is internally coated with oxygen-enriched oil releasing reactive oxygen species and is free from active pharmaceutical ingredients. It is intended, among other indications, for the use in surgical wounds after oncological breast surgery, breast reconstruction and cosmetic breast surgery. In two studies, a total of 140 patients (surgical wounds after breast augmentation-mastopexy, mammary lesions) were treated successfully with NovoX® Cup and no product-related adverse events were reported.The claimed advantages sound promising but an advantage compared to established wound dressings such as sterile strips or tapes has still to be investigated.

The aim of the following study is to compare the outcomes (postoperative complications, scar quality and patients' satisfaction) of breast reduction and application of the wound dressing NovoX® Cup in comparison to already established wound closure systems 2 weeks and 3 months after surgery.

DETAILED DESCRIPTION:
A prospective intra-individually controlled cohort study.

One breast will be chosen (left or right) to be treated with the NovoX®-Cup.

The other breast will serve as the "standard of care" control.

Randomization within this clinical investigation will be done intra-individually in a 1:1 ratio.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Female patients 18 years and older
* Patient able to give informed consent
* Patients undergoing bilateral breast reduction

Exclusion Criteria:

* Absent informed consent
* Patients from protected groups and those who are not personally able to give consent.
* Patients younger than 18 years
* Pregnancy (pregnancy test before enrollment) and breastfeeding women
* Former radiation of the breast(s)
* Former surgery at the operation site
* Skin abnormalities in the operation area (e.g. burn scars)
* Participation in other clinical trials during this study
* Active malignant disease
* Breast cancer history
* Radiation or chemotherapy during the study period or up to 6 months before possible enrollment
* Immune disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female patients undergoing elective bilateral breast reduction surgery.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-07-25 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Scar quality (Vancouver Scar Scale, VSS) | 2 weeks and 3 months after surgery.
  scar quality measured through VSS scale (total scores 0 to 13), higher scores indicate worse scar outcome
Scar quality (Patient and Observer Scar Assessment Scale, POSAS) | 2 weeks and 3 months after surgery.
  scar quality measured through POSAS scale (total scores 6 to 60), higher scores indicate worse scar outcome
Wound healing disorder | 2-weeks and 3 months post-surgery
  occurrence of wound healing disorders (yes/no)

SECONDARY OUTCOMES:
Pain (Numerical Scale Rating NRS) | before surgery, 2-weeks and 3 months post-surgery
  Pain evaluated with Numerical Scale Rating (NRS score 0 to 10) higher score indicates worse pain
Surgical Complications (Clavien-Dindo-Classification CDC) | 3 months post-surgery
  Clavien-Dindo-Classification (CDC grade I to V) of surgical complications, higher grade indicates higher severity of the complications
Breast-Q® Outcome | before surgery, 2 weeks and 3 months post-surgery
  Breast-Q® questionnaire satisfaction with outcome (scores 0 - 100 for each breast), higher score indicates greater satisfaction
Breast-Q® breasts | before surgery, 2 weeks and 3 months post-surgery
  Breast-Q® questionnaire satisfaction with breasts (scores 0 - 100 for each breast), higher score indicates greater satisfaction
Breast-Q® nipples | before surgery, 2 weeks and 3 months post-surgery
  Breast-Q® questionnaire satisfaction with nipples (scores 0 - 100 for each breast), higher score indicates greater satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Lars-Peter Kamolz, Prof., Principal Investigator — Medical University of Graz, Austria
Locations (1):
- Division of Plastic, Aesthetic & Reconstructive Surgery, Department of Surgery, Medical University of Graz, Graz, Austria

IPD SHARING:
Plan to Share IPD: No